CLINICAL TRIAL: NCT01231854
Title: Ciclosporin Versus Alitretinoin for Severe Atopic Hand Dermatitis. A Randomized Controlled Investigator-initiated Double-blind Trial.
Brief Title: Ciclosporin Versus Alitretinoin for Severe Atopic Hand Dermatitis.
Acronym: TocyDD
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: delayed start of the trial, both treatment options already have market authorizations, study medication expired
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TUD-TOCYDD-044; 2009-017520-88 (EudraCT Number)
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-06

CONDITIONS: Atopic Dermatitis
Keywords: atopic hand dermatitis; Chronic hand dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Cyclosporine; Alitretinoin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ciclosporingroup (Active Comparator)
  Interventions: Drug: Ciclosporin
- Alitretinoingroup (Active Comparator)
  Interventions: Drug: Alitretinoin

INTERVENTIONS:
Drug: Ciclosporin — In accordance with the current guideline concerning the use of ciclosporin in dermatology and the current guideline management of hand eczema the daily oral dosage of ciclosporin microemulsion is 2.7 to 4.0 mg/kg bodyweight (half of the total daily dosage will be administered in the morning and in the evening). To enable both body-weight adjusted treatment and double-blind treatment patients will be allocated to 2 different dosages depending on their body weight (50-74.9 kg: daily dosage 200 mg; 75-100 kg: daily dosage 300 mg).
  Other Names: Immunosporin
  Arms: Ciclosporingroup
Drug: Alitretinoin — In accordance with the current guideline management of hand eczema alitretinoin will be administered orally in a constant daily dosage of 30 mg.
  Other Names: Toctino
  Arms: Alitretinoingroup

SUMMARY:
The purpose of this study is to investigate the comparative efficacy, safety and efficiency of ciclosporin microemulsion and alitretinoin in adults with severe atopic hand dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female Patients age > 18 years and ≤ 75 years
* Body weight 50 to 100 kg
* Chronic hand dermatitis (duration > 6 months)
* Atopic constitution according to

  * Erlanger Atopiescore1 and/or
  * positive personal history for atopic eczema, allergic rhinitis, allergic asthma and/or
  * elevated serum IgE
* Severe hand dermatitis not responding to treatment with potent topical steroids for at least 4 weeks within the past 6 months due to IGA
* Written informed consent

Exclusion Criteria:

* Participation in other clinical trial within past 4 weeks
* Pregnancy/breastfeeding
* Women within reproductive age except those women who fulfil at least one of the following criteria throughout the total study and until at least 5 weeks after active study treatment in case of early study termination:
* post-menopausal women (12 months physiological amenorrhoea or 6 months amenorrhoea with serum FSH level > 40 mlU/ml),
* postoperative (6 weeks after bilateral ovariectomy with or without hysterectomy)
* Regular and proper use of at least two methods of contraception, including at least one method of contraception with a failure rate <1% per year (eg, implants, depot preparations, oral contraceptives, IUD).
* vasectomy of the partner.
* Women within reproductive age, who do not meet all of the following criteria throughout the whole study or - in case of early study termination - up to 5 weeks after active therapy:
* The patient understands the teratogenic risk associated with taking the study medication.
* The patient understands the need for strict monthly monitoring, the need for a reliable, continuous contraception and the need for regular pregnancy tests throughout the study and - in case of early study termination - up to 5 weeks of active therapy.
* The patient is able to adequately and reliably apply methods of contraception.
* The patient is informed about the possible consequences of pregnancy and knows that she must immediately contact her physician in case of suspected pregnancy.
* The patient gives informed consent about knowing the potential risks and necessary measures to avoid pregnancy.
* Blood and/or plasma donation during the whole study period. In case of early study termination blood and plasma donation is not allowed until 1 month after the end of active study treatment
* UV-therapy within past 3 months
* Concurrent photo-and / or photochemotherapy
* Known Hypersensitivity / Intolerance against ciclosporin, alitretinoin or any other ingredients of Immunosporin® or Toctino®
* Known Allergy against peanuts or soya
* Known Hereditary fructose intolerance
* Acute and/or uncontrolled chronic infectious disease
* Known Congenital or acquired immune deficiency
* Malignant tumor (past or present)
* Uncontrolled arterial hypertension (RR systolic ≥ 160 mm Hg and/or RR diastolic≥ 90 mm Hg despite anti-hypertensive treatment)
* Renal insufficiency (Serum creatinine above normal range)
* Liver insufficiency (CHILD ≥ Stadium B)
* Not sufficiently controlled hyperlipidemia (LDL/HDL ratio > 4 despite medical treatment)
* Clinically significant thyroid hypofunction
* Known Hypervitaminosis A
* Concurrent supplementation of vitamin A or treatment with other retinoids
* Concurrent tetracycline therapy
* Concurrent therapy with St. John's wort ("Johanniskraut")
* Known genetic diseases causing increased UV light sensitivity such as Xeroderma pigmentosum, Cockayne-syndrome, Bloom syndrome
* Known Drug- and/or alcohol abuse
* Known significant psychiatric morbidity

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with complete or almost complete clearance according to the Investigator Global Assessment (IGA) within 24-week active therapy in both groups.

SECONDARY OUTCOMES:
Time to complete or almost complete clearance according to IGA in both groups
Proportion of patients with complete or almost complete clearance according to the Patients Global Assessment (PGA) within 12 weeks and 24 weeks of active therapy
Mean relative change in objective disease severity (HECSI) between baseline and week 4, 8, 12, 16, 20, 24 in both groups
Mean relative change in quality of life (Skindex 17) between baseline and week 24 in both groups
Cost-effectiveness of the studied treatment options (cost / QALY gained; assessed by means of the (EQ-5D)
Mean relative change in work productivity (assessed by means of the work limitations questionnaire (WLQ) in both groups
Mean utilization of topical steroids within the follow-up period in both groups
Patient satisfaction with treatment in both groups (assessed using a 100mm VAS Scale)
Proportion of patients with relapse (≥ 75% of baseline HECSI) within 24-week follow-up after previous complete/almost complete clearance
In patients with atopic dermatitis on the body: measured percentage of patients with at least 50% improvement in disease severity with the active therapy using the SCORAD.
Tolerability and safety in both study groups

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsklinikum Carl Gustav Carus an der TU Dresden, Dresden, Saxony, Germany